CLINICAL TRIAL: NCT05763901
Title: Evaluation of Motor Control During Developmental Age in Young Patients With Paramorphisms and Dysmorphisms Using Inertial Measurement Units
Brief Title: IMU-based Assessment of Motor Control in a Population of Young Subjects With Paramorphisms and Dysmorphisms
Acronym: MOTOR-CHILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0004188
Record Dates: First submitted 2022-07-14; First posted 2023-03-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Genu Varum; Genu Valgus; Flat Feet; Cavus Foot; Scoliosis Idiopathic; Varus; Talipes; Valgus, Talipes; Laxity of Ligament; Hyperlordosis; Hyperkyphosis; Angular Limb Deformity
MeSH Terms: conditions — Genu Varum; Genu Valgum; Flatfoot; Talipes Cavus; Clubfoot; Joint Instability; Swayback; Kyphosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paramorphisms/dysmorphisms of spine and/or lower limbs (Experimental): Only one arm of patients assessed for motor competence and balance without controls
  Interventions: Diagnostic Test: Clinical tests and motor control evaluation using Inertial Measurement Units

INTERVENTIONS:
Diagnostic Test: Clinical tests and motor control evaluation using Inertial Measurement Units — Each patient is evaluated using clinical tests (Movement ABC2, Test of Motor Competence), a screening questionnaire (DCD-Q), and wearable Inertial Measurement Units to assess balance and motor control during a Natural Walking and Tandem Walking test.

SUMMARY:
While various complex pathologies of the developmental age, such as Infantile Cerebral Palsy or Neuromuscular Diseases, are notoriously considered causes of alteration of locomotor development, it is scarcely known whether conditions much more frequent in the pediatric population, the so-called "Paramorphisms or Dysmorphisms", may be associated with more or less noticeable changes in locomotor development.

On a few studies, flat feet and hyperlaxity has been correlated with a motor control delay or poorer motor performance, based on complex clinical tests or on stereophotogrammetry movement analysis.

Although promising, these preliminary studies, in addition to not providing information on the possible influence of other paramorphisms, such as varus and valgus of the knees, do not provide conclusive indications.

The aim of this study is to investigate, through clinical tests and wearable inertial units, the motor control of a pediatric population affected by Paramorphisms or Dysmorphisms and to compare them with a population of healthy controls, matched by age, taken from the recently developed control data set from Bisi and Stagni.

ELIGIBILITY:
Inclusion Criteria:

* Born at term
* Without known delay in motor development
* Finding of one or more paramorphisms or dysmorphisms of the developmental age (flat or cavus foot, valgus or varus talipes, valgus or varus knee, scoliotic attitude or scoliosis, hyperkyphosis or hyperlordosis, generalized or focused hyperlaxity, heterometry of the AAII, torsional defects AAII)

Exclusion Criteria:

* Preterm birth
* Diagnosis of pathologies compromising motor control (Infantile Cerebral Palsy, Neuromuscular Diseases, Spina Bifida, Arthrogryposis, Genetic Syndromes)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluation and measurement of balance | Baseline
  Evaluation of balance using clinical tests ( Movement ABC2).
Evaluation and measurement motor competence | Baseline
  Evaluation of motor competence using clinical tests (Test of Motor Competence, ).
Measurement of balance | Baseline
  Measurement of balance assessing synchronicity from data obtained with Inertial Measurement Units.
Measurement of motor competence | Baseline
  Measurement motor competence assessing automaticity from data obtained with Inertial Measurement Units.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS-Istituto Ortopedico Rizzoli, Bologna, Italy